CLINICAL TRIAL: NCT04554290
Title: Giant Cell Arteritis and Differential Diagnoses Associated With Positive Temporal Artery Biopsy: a Monocentric Retrospective Study
Brief Title: Giant Cell Arteritis and Differential Diagnoses Associated With Positive Temporal Artery Biopsy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Thomas MOULINET, MD, Central Hospital, Nancy, France
Other Study IDs: 2020PI061
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Giant Cell Arteritis; Vasculitis
Keywords: giant cell arteritis; temporal artery biopsy; vasculitis
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- positive temporal artery biopsy: all adult patients with significant inflammation shown on temporal artery biopsy
  Interventions: Diagnostic Test: temporal artery biopsy

INTERVENTIONS:
Diagnostic Test: temporal artery biopsy — description of temporal artery biopsy features, and its correlation with diagnosis of giant cell arteritis or other differential diagnoses.

SUMMARY:
Temporal artery biopsy is a useful tool helping to the diagnosis of giant cell arteritis. However, other diagnoses might be associated with abnormal temporal artery biopsy. The purpose of this study is to describe the frequency of giant cell arteritis differential diagnoses with positive temporal artery biopsy.

ELIGIBILITY:
Inclusion Criteria:

* positive artery biopsy between january 1st 2000 and july 25th 2019

Exclusion Criteria:

* orther vascular biopsy than temporal artery biospy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with significant inflammation on temporal artery biospy, with a final diagnosis of giant cell arteritis or an other diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
percentage of giant cell arteritis and differential diagnoses | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital, Nancy, Lorraine, France

REFERENCES:
- [Result] Pontille F, Decker P, Gauchotte G, Jaussaud R, Moulinet T. Diagnoses associated with temporal arteritis. Eur J Intern Med. 2023 Nov;117:140-143. doi: 10.1016/j.ejim.2023.08.010. Epub 2023 Aug 14. No abstract available. PMID 37586985